CLINICAL TRIAL: NCT06053814
Title: A Phase 1/2, First in Human, Multiple-dose, 2-part Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of NS-050/NCNP-03 in Boys With Duchenne Muscular Dystrophy (DMD)
Brief Title: NS-050/NCNP-03 in Boys With DMD (Meteor50)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NS Pharma, Inc. (Industry)
Collaborators: Nippon Shinyaku Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NS-050/NCNP-03-101
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: NS-050/NCNP-03 (Experimental): Participants will be randomized and receive NS-050/NCNP-03 intravenous (IV) infusions once weekly for 2 weeks at each of MAD levels (1.95, 5, 10, 20, 40, and 80 mg/kg).
  Interventions: Drug: NS-050/NCNP-03
- Part 1: Placebo (Placebo Comparator): Participants will be randomized and receive NS-050/NCNP-03 placebo-matching IV infusions once weekly for 2 weeks at each of MAD levels.
  Interventions: Drug: Placebo
- Part 2: NS-050/NCNP-03 (Experimental): Participants will receive NS-050/NCNP-03 IV infusions once weekly for 24 weeks at the dosage selected by the Data and Safety Monitoring Board (DSMB) at the conclusion of Part 1.
  Interventions: Drug: NS-050/NCNP-03

INTERVENTIONS:
Drug: NS-050/NCNP-03 — NS-050/NCNP-03 solution for IV infusion.
  Arms: Part 1: NS-050/NCNP-03; Part 2: NS-050/NCNP-03
Drug: Placebo — NS-050/NCNP-03 placebo-matching solution for IV infusion.
  Arms: Part 1: Placebo

SUMMARY:
This is a Phase 1/2 study of Multiple-Ascending Dose (MAD) levels for 12 weeks of treatment followed by 24 weeks of open-label treatment with a selected dose of NS-050/NCNP-03 administered once weekly to ambulant boys with DMD, who have a DMD exon deletion amenable to exon 50 skipping.

ELIGIBILITY:
Inclusion Criteria:

* Male ≥ 4 years and <15 years of age;
* Confirmed DMD exon deletion in the dystrophin gene that is amenable to skipping of exon 50 to restore the dystrophin mRNA reading frame;
* Able to walk independently without assistive devices;
* Able to complete the TTSTAND without assistance in <20 seconds;
* Stable dose of glucocorticoid for at least 3 months and the dose is expected to remain on a stable dose for the duration of the study.

Other inclusion criteria may apply.

Exclusion Criteria:

* Evidence of symptomatic cardiomyopathy;
* Current or previous treatment with anabolic steroids (e.g., oxendolone, oxandrolone) or products containing resveratrol or adenosine triphosphate within 3 months prior to first dose of study drug;
* Currently taking another investigational drug or has taken another investigational drug within 3 months prior to the first dose of study drug;
* Surgery within the 3 months prior to the first dose of study drug or planned during the study duration;
* Having taken any gene therapy.

Other exclusion criteria may apply.

Ages: 4 Years to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Part 1: Overall Summary of Treatment-emergent Adverse Events (TEAEs) | Baseline up to Week 24
  TEAEs will be summarized both at the patient level for number of TEAEs, highest severity, relationship, action, and outcome, and at the TEAE level (summarizing events) by system organ class (SOC) and preferred term (PT) as well as severity, relationship, action, and outcome.
  The most recent version of the Medical Dictionary for Regulatory Activities (MedDRA) will be used for coding TEAEs.
Part 1: Area Under the Plasma Concentration Versus Time Curve (AUC) of NS-050/NCNP-03 | Day 1 (1st dose) for each dose level
  Blood samples will be collected at the designated time frame. Pharmacokinetic (PK) parameters of NS-050/NCNP-03 will be calculated using non-compartmental methods.
Part 1: Amount of Drug Excreted in Urine of NS-050/NCNP-03 | Day 1 (1st dose) for each dose level
  Urine samples will be collected at the designated time frame. PK parameters of NS-050/NCNP-03 will be calculated using non-compartmental methods.
Part 2: Change from baseline in skeletal muscle dystrophin protein by immunoblot (Western blot) | Baseline, Week25

SECONDARY OUTCOMES:
Part 2: Change from baseline in skeletal muscle dystrophin protein by mass spectrometry | Baseline, Week25
Part 2: Change from baseline in skeletal muscle dystrophin protein levels by immunofluorescence staining | Baseline, Week25
Part 2: Change from baseline in percentage of exon 50-skipped mRNA of skeletal muscle dystrophin | Baseline, Week25
Part 2: North Star Ambulatory Assessment (NSAA) score | Baseline, Week13, Week25
  The NSAA is a functional scale devised for use in ambulant children with Duchenne muscular dystrophy (DMD). It consists of 17 activities graded 0 (unable to perform), 1 (performs with modifications), 2 (normal movement). It assesses abilities necessary to remain ambulant that have been found to progressively deteriorate in untreated DMD patients, as well as in other muscular dystrophies such as Becker Muscular Dystrophy. NSAA Total Score ranges from 0 to 34, with a score of 34 implying normal function.
Part 2: Time to Stand (TTSTAND) | Baseline, Week13, Week25
Part 2: Time to Run/Walk 10 Meters (TTRW) | Baseline, Week13, Week25
Part 2: Time to Climb 4 Stairs (TTCLIMB) | Baseline, Week13, Week25
Part 2: Total distance of 6 Minute Walk Test (6MWT) | Baseline, Week13, Week25
Part 2: Muscle strength measured by Quantitative Muscle Testing (QMT) | Baseline, Week13, Week25
Part 2: Grip/Pinch Strength | Baseline, Week13, Week25
Part 2: Performance of Upper Limb (PUL) 2.0. score | Baseline, Week13, Week25
  The PUL 2.0 provides both a total score and sub-scores for the 3 domains (shoulder, middle, and distal) that in DMD are progressively involved with a proximal to distal gradient. The PUL includes 22 items with an entry item to define the starting functional level. The 22 items are subdivided into the high level shoulder dimension (6 items), middle level elbow dimension (9 items), and distal wrist and hand dimension (7 items). For weaker patients, a low score on the entry item (0 2) means high level items do not need to be performed. Scoring options vary across the scale between 0-1 and 0-2 according to performance. Each dimension can be scored separately with a maximum score of 12 for the high level shoulder dimension, 17 for the middle level elbow dimension, and 13 for the distal wrist and hand dimension. A total score can be achieved by adding the 3 level scores (maximum total score of 42).

CONTACTS AND LOCATIONS:
Locations (18):
- United States (6):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- Canada (3):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - London Health Sciences Centre, London, Ontario
- Japan (4):
  - National Hospital Organization Nagara Medical Center, Nagara, Gifu
  - Hyogo Medical University Hospital, Nishinomiya, Hyōgo
  - NHO Osaka Toneyama Medical Center, Toyonaka, Osaka
  - National Center of Neurology and Psychiatry, Kodaira, Tokyo
- South Korea (2):
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Seoul National University Hospital, Seoul
- Turkey (Türkiye) (3):
  - Ankara Bilkent City Hospital, Ankara
  - Istanbul University, Istanbul
  - Yeditepe University Kosuyolu Hospital, Istanbul